CLINICAL TRIAL: NCT06818162
Title: MULTICENTER ULNAR NERVE ULTRASONOGRAPHIC and NEUROPHYSIOLOGICAL STUDY: NORMATIVE DATA COLLECTION
Acronym: US-ULN
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Ubaldo Del Carro, MD Responsible of the Neurophysiology Unit and Director of the Intraoperative Monitoring., IRCCS San Raffaele
Other Study IDs: US-ULN
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Collecting Normative Data of Ulnar Nerve CSA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: normative data — Ultra sonography of ulnar nerve along its course to obtain normative values for the CSA

SUMMARY:
The study population will include a total of 500 subjects, selected from outpatients accessing the Neurophysiology Service for a neurophysiological study of the upper limbs. Only those whose neurophysiological examination results negative for Peripheral Nervous System pathology (i.e., negative electroneurography and electromyography according to AANEM guidelines) will be recruited. The subjects will be enrolled in 22 centers distributed throughout Italy, with our center planning to recruit 50 subjects.

The diagnostic procedures include electroneurography and electromyography, which are standard clinical practice. Ultrasound (ultrasonographic study) is not an experimental technique but is considered an additional procedure specifically included in the study protocol.

The primary objective of the study is to establish normative values for the CSA of the ulnar nerve and assess the reliability of the measurement through inter-operator comparison (between a physician and a neurophysiology technician). Therefore, during an evaluation lasting approximately 30-60 minutes, the enrolled subjects will undergo an electroneurographic/electromyographic and ultrasound study of the ulnar nerve. The latter will be performed by two independent operators (a physician and a neurophysiology technician).

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old EMG/ENG completely negative for pathologies of the peripheral nervous system (ENG and EMG negative according to the regulatory data of each single Center) Signature of the informed consent

Exclusion Criteria:

* Diabetes, Hepatitis, Renal Failure History of NPL or previous CT Previous pathologies of the peripheral nervous system Previous trauma to the limb in question Positive familiarity for neuromuscular disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with indication to perform an EMG/ENG for upper limb which fulfill inclusion/exclusion criteria
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
CSA Normative value | single evaluation
  CSA Normative value of ulnar nerve at the wrist, below, at, above the elbow, at Axilla, CSA above elbow/CSA below elbow ratio